CLINICAL TRIAL: NCT01022840
Title: The Opioid Sparing Effect of Minimal Dose S-Ketamine Applied as a Coanalgesic During the Perioperative Period - An Active Placebo-Controlled, Double Blinded, Randomized Clinical Trial (МiniKet)
Brief Title: The Preemptive Analgetic Potency of Low Dose S-Ketamine
Acronym: Miniket
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Andreas Sandner-Kiesling , MD, Univ. Prof. Dr., Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 180808
Record Dates: First submitted 2009-11-21; First posted 2009-12-01 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Esketamine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo as saline solution
  Interventions: Other: Placebo Comparison
- Low dose (Experimental): S-Ketamine
  Interventions: Drug: S-Ketamine
- High dose (Active Comparator)
  Interventions: Drug: S-Ketamine

INTERVENTIONS:
Drug: S-Ketamine — drug
  Other Names: Ketanest
  Arms: High dose; Low dose
Other: Placebo Comparison — saline control
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The primary hypothesis is improved postoperative analgetic quality using S-Ketamine, particularly in patients suffering from chronic pain.

DETAILED DESCRIPTION:
The investigators are dealing mainly with the finding of the right dosage for the optimal safety and efficacy of S-Ketamine, but also discovering new possible areas of investigation (e.g. anti-depressive effect, anti-neuropathic effect).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for major abdominal surgery
* Suitable for PCA
* Cardio-vascular stable
* Age: 18+
* Between 50-120kg BW
* ASA 1-3
* Good Compliance for pain monitoring

Exclusion Criteria:

* Allergy to S-Ketamine
* Severe liver or kidney dysfunction
* Severe coronary disease
* Pregnancy
* Present or past psychotic disorders
* Addiction to alcohol or opioids
* Poor compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-02; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
postoperative opioid consumption | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mischa Wejbora, MD, Principal Investigator — Med. U Graz
Locations (3):
- Austria (3):
  - Medical University Graz, Graz, Styria
  - Medical University of Graz, Graz, Styria
  - Medical University of Graz, Graz